CLINICAL TRIAL: NCT00327145
Title: A Double-blind, Randomized, Multicenter Study to Evaluate the Effectiveness of the Combination of Valsartan & Amlodipine in Hypertensive Patients Not Controlled on Monotherapy
Brief Title: A Study to Evaluate the Combination of Valsartan and Amlodipine in Hypertensive Patients Not Controlled on Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAA489A2401
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: HCTZ; hypertension; valsartan; amlodipine
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide; Amlodipine

INTERVENTIONS:
Drug: valsartan
Drug: hydrochlorothiazide
Drug: amlodipine

SUMMARY:
This study is designed to provide additional efficacy and safety data for a treatment strategy based on the combination valsartan with amlodipine in hypertensive patients previously treated with monotherapy and remaining uncontrolled. A naturalistic approach will be taken comparing two different doses, i.e. 160mg of valsartan with amlodipine 5mg and 10mg with possible addition of HCTZ

ELIGIBILITY:
Inclusion criteria

* Male or female patients ≥18 years of age
* Non-diabetic patients must have MSSBP of ≥140 mmHg and/or MSDBP ≥90 mmHg at Visits 1 and 2. Diabetic patients must have MSSBP ≥130 mmHg and/or MSDBP ≥80 mmHg at Visits 1 and 2
* Patients treated with monotherapy at a dose considered as adequate by the investigator for a minimum of two months prior to Visit 1

Exclusion criteria

* Known or suspected contraindications, including history of allergy to ARBs, CCB, thiazides or to drugs with similar chemical structure.
* MSSBP ≥180 mmHg and/or MSDBP ≥110 mmHg (MSSBP ≥160 mmHg and/or MSDBP ≥100 mmHg for diabetic patients) at any time between Visit 1 and Visit 2.
* Evidence of a secondary form of hypertension, to include coarctation of the aorta, primary hyperaldosteronism, renal artery stenosis, or pheochromocytoma.
* Known Keith-Wagener grade III or IV hypertensive retinopathy.
* Other exclusion criteria apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 894 (Actual)
Dates: Start 2006-03; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure less than 140/90 mmHg in non diabetic patients or blood pressure less than 130/80 mmHg in diabetic patients after 16 weeks

SECONDARY OUTCOMES:
Blood pressure less than 140/90 mmHg in non diabetic patients or blood pressure less than 130/80 mmHg in diabetic patients after 8 weeks.
Blood pressure less than 140/90 mmHg in non diabetic patients or blood pressure less than 130/80 mmHg in diabetic patients after 4, 12, and 16 weeks.
Change from baseline diastolic and systolic blood pressure measurements after 4, 8, 12, and 16 weeks
Diastolic blood pressure less than 90 mmHg in non-diabetic patients and diastolic blood pressure less than 80 mmHg in diabetic patients after 4, 8, 12, and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Allemann Y, Fraile B, Lambert M, Barbier M, Ferber P, Izzo JL Jr. Efficacy of the combination of amlodipine and valsartan in patients with hypertension uncontrolled with previous monotherapy: the Exforge in Failure after Single Therapy (EX-FAST) study. J Clin Hypertens (Greenwich). 2008 Mar;10(3):185-94. doi: 10.1111/j.1751-7176.2008.07516.x. PMID 18326958